CLINICAL TRIAL: NCT06116565
Title: An Multi-center, Open-label, Single-arm Phase 2 Study to Evaluate the Long-term Safety and Efficacy of CM310 in Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study of CM310 in Subjects With Moderate-to-Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310-101116
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental)
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310, subcutaneous injection

SUMMARY:
This is a multi-center, open-label phase 2 study to evaluate the long-term safety and efficacy of CM310 in subjects with moderate-to-severe atopic dermatitis.

DETAILED DESCRIPTION:
The study consists of an screening period, treatment period, and safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study and voluntarily sign a written informed consent form (ICF).
* Age ≥ 18 and ≤ 75 years old.
* With Atopic Dermatitis.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Concurrent disease/status which may potentially affect the efficacy/safety judgement.
* Major surgeries are planned during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | up to Week 60
  Incidence of adverse events (AEs).